CLINICAL TRIAL: NCT05421923
Title: A Phase I Bridging Study to Evaluate the PK, PD, Safety and Tolerability of SR1375 in Healthy Subjects
Brief Title: The Pharmacokinetics (PK), Pharmacodynamics(PD), Safety, Tolerability of SR1375 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai SIMR Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SR1375-102
Record Dates: First submitted 2022-06-10; First posted 2022-06-16 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SR1375 capsules (Experimental): Ascending single and multiple doses of SR1375 orally
  Interventions: Drug: SR1375 capsules
- Placebo (Placebo Comparator): Ascending single and multiple doses of SR1375 placebo orally
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SR1375 capsules — Ascending single and multiple doses of SR1375 orally
  Arms: SR1375 capsules
Other: Placebo — Ascending single and multiple doses of Placebo orally
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase I bridging study to evaluate the PK, PD, safety and tolerability of SR1375 in healthy subjects.

DETAILED DESCRIPTION:
The study is a Phase I study to evaluate the PK, PD, safety, and tolerability of SR1375 in healthy volunteers. The study will include 3 single-ascending-dose (SAD) cohorts and 1 multiple-dose cohorts (Part A and part B respectively), a total of 4 cohorts, and each cohort includes 3 stages: screening and baseline, treatment and safety monitoring, and safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females who are 18 to 45 years of age.
2. Based on medical history, physical examination, laboratory examination, chest CT scan, abdominal B-ultrasound, vital signs and ECG, the investigator considered that the results were normal or abnormal but no clinical significance.
3. Bodyweight of male > 50 kg, Bodyweight of female > 45 kg and body mass index (BMI) between 18 and 28 kg/m2.
4. Male subjects must agree to use a highly effective contraceptive method from signing the consent form until at least 90 days after the last dose of study drug, and must be willing not to donate sperm.
5. Healthy female volunteers must be:

   i. Of non-childbearing potential(with a documented tubal ligation, bilateral salpingectomy, hysterectomy, or menopause for more than 1 year) ii. Of childbearing potential, must have a negative pregnancy test at the screening visit (blood test), must agree to use a highly effective contraceptive method from signing the consent form until at least 30 days after the last dose of study drug.
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. History of hypercoagulable state or history of thrombosis.
2. Current or chronic history of liver disease or known hepatic or biliary abnormalities.
3. History of sensitivity to any of the investigational medicinal products (IMPs), or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates participation.
4. History of asthma (excluding resolved childhood asthma), severe allergic responses.
5. History of significant drug abuse within one year of screening.
6. Except for topical (no significant systemic exposure) permitted, use of the following combination agents will be excluded:

   1. Use of prescription drugs within 14 days prior to initial administration, or within 7 days or five half-lives of the medication (whichever is longer) prior to the first study drug administration, except occasional use of paracetamol (up to a maximum of 2000 mg per day of paracetamol and per local or national abelling).
   2. Use the health supplement 7 days or 5 half-life before the first administration of the investigational drug.
   3. Use of depot injection or subcutaneous implantation drugs within 3 months prior to the first study drug administration.
   4. Received vaccine within 1 month prior to the first administration of the investigational drug.
7. A positive Hepatitis B surface antigen, positive Hepatitis C antibody and positive test for human immunodeficiency virus (HIV) antibody or treponema pallidum antibody.
8. A positive drug/alcohol result.
9. History of regular alcohol consumption within 6 months of screening defined as:

   an average weekly intake of >14 units (1 unit of alcohol ≈360 mL beer or 45 mL 40% alcohol spirits or 150 mL wine), or abstain from alcohol during the study.
10. Within 6 months of screening, smoking more than 5 cigarettes(including e- cigarettes).
11. Donation or lost in excess of 400 mL of blood within 2 months of Day 1 or donation of plasma within 14 days of Day 1.
12. The subject has participated in a clinical trial within 3 months of receiving IMP.
13. Unable to refrain from consumption of Seville oranges, grapefruit or grapefruit juice within 24h prior to the first dose of IMP until the Safety Follow-up visit.
14. Breast-feeding and/or lactating subject.
15. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Cmax | On scheduled intervals from Day 1 up to Day 54
  Peak plasma concentration
Tmax | On scheduled intervals from Day 1 up to Day 54
  Time of peak plasma concentration
AUC | On scheduled intervals from Day 1 up to Day 54
  Area under the plasma concentration-time curve
CL/F | On scheduled intervals from Day 1 up to Day 54
  Apparent oral clearance
t1/2 | On scheduled intervals from Day 1 up to Day 54
  Terminal half-life
Rac | On scheduled intervals from Day 1 up to Day 54
  Accumulation ratio

SECONDARY OUTCOMES:
The frequency and severity of AEs in healthy volunteers administrated with single and repeated oral doses of SR1375 capsules | On scheduled intervals from Day 1 up to Day 54
  AE: Adverse Event
PAF-AH | On scheduled intervals from Day 1 up to Day 54
  Platelet activating factor acetylhydrolase

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Jing, Principal Investigator — Phase I clinical laboratory of Huashan Hospital
Locations (1):
- Phase I clinical laboratory of Huashan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No